CLINICAL TRIAL: NCT03218189
Title: Differences Between Essential Medicines Lists in 135 Countries and the World Health Organization's Model List of Essential Medicines
Brief Title: Differences Between Essential Medicines Lists in 135 Countries and Model List of Essential Medicines
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-308
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Formularies
Keywords: Essential medicines lists

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Country characteristics — Observational study of country characteristics

SUMMARY:
The World Health Organization (WHO) has developed a model list of more than 400 medicines and recommends that each country adapt the list to its own circumstances. More than 100 countries have developed essential medicines lists.

Some countries have essential medicines lists that are very similar to the WHO's model list and other countries have lists that are very different from the WHO's model list. Differences between the WHO list and country lists could be explained by features of the country including population demographics, disease prevalence, Gross Domestic Product (GDP), and healthcare system organization. Other factors such as the influence of particular individuals or organizations may also explain differences between countries.

The purpose of this project is to compare the essential medicines lists developed by countries with the WHO's model list and to identify attributes of countries that are associated with differences from the WHO list. Predictors such as region, population, life expectancy, infant mortality rate, GDP per capita, health expenditure per capita, inequality, and the corruption perception index will be considered.

DETAILED DESCRIPTION:
Statistical analysis plan for objective 3 (relationship between the total number of differences and country features)

Plots will be generated to show the relationships between variables. Correlation coefficients will be calculated where appropriate. Two separate multivariate models will be fit to the data for outcomes 2a and 2b [continuous, between 1 and 500]. A similar model will be fit the total number of differences. The analytical method will be determined by the data and may be liner regression.

Predictors:

Region-Categorical (6)

Population-Continuous

Life expectancy-Continuous

Infant mortality rate-Continuous

GDP per capita-Continuous

Health expenditure per capita

Inequality-Continuous

Corruption Perception Index-Continuous

ELIGIBILITY:
Inclusion Criteria:

* Countries that have an essential medicines list, and Canada

Exclusion Criteria:

* countries that do not have an essential medicines list that is available online

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Countries that have an essential medicines list are included in the study
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Total number of differences between the WHO model list of essential medicines and the essential medicines list in each country | 1 year
  The total number of differences between the WHO model list of essential medicines and the essential medicines list in each country is comprised of:
  1. number of WHO model list medicines not on country list including the number of substitutions within class (i.e. a medicine on WHO list not on country's list but a similar agent in the same class is on the country's list); and the
  2. number of medicines on the country list but not on the WHO model list.

SECONDARY OUTCOMES:
Medications that are on the WHO list but not on the country list | 1 year
Medications that are on the country list but not on the WHO list | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
At the time of publication, we will publicly post a table with the country characteristics and the outcomes
Time Frame: At the time of publication.
Access Criteria: Publicly posted.